CLINICAL TRIAL: NCT06291558
Title: A Comparison of Exercise Education Outcomes Based on Nicotine Addiction Levels in Smoking Students
Brief Title: Exercise Training for Smoking Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Fulya Demirhan, Research Assistant, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P202200027
Record Dates: First submitted 2024-02-09; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Nicotine Dependence; Smoking; Physical Inactivity; Depression
Keywords: resistance exercise; respiratory exercise; nicotine addiction; respiratory function test; telehealth
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Sedentary Behavior; Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be informed that the study was carried out for scientific purposes and the information will not be shared with third parties. Randomization of exercise groups will be performed according to the closed envelope procedure. The student who selects one of the envelopes with the names of the 3 groups will be included in the group written in the envelope he selected. Information about other groups will not be shared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face to face Exercise Group (Experimental): In the face-to-face exercise group called Group 1, students will implement an exercise program of respiratory exercises and resistance exercises with the physiotherapist. Exercises will be held for 8 weeks
  Interventions: Other: Exercise
- Telehealth Exercise Group (Experimental): In the online (telehealth) exercise group, group 2 will be applied by the students with the help of the physiotherapist. Exercises will be held for 8 weeks
  Interventions: Other: Exercise
- Control Group (No Intervention): In the control group called Group 3, students will not be given any exercise program.

INTERVENTIONS:
Other: Exercise — The first 5 minutes of heating in the exercise program are planned to be implemented for 8 weeks, and the last 5 minutes are a cooling period. In the exercise program, which is planned to last 40 minutes in total, respiratory exercises will be applied to heating and cooling peryotes. As respiratory exercise, diaphragmatic respiratory exercise will be applied to heating and cooling peryots with 5 repetitions. Elastic resistant bands (Therand) will be used in resistant exercise training that will last for 30 minutes. The participants will be started to work with the resistance that they can do 10 again but cannot reach 14 repetitions. Elastic resistant bands are shoulder flexion, shoulder extension, shoulder ablution, shoulder horizontal abduction, elbow extension, hip ablution, hip flexion, and hip exercise. These exercises will be held once a week, 10 repetitions, 2 sets, for 8 weeks.
  Arms: Face to face Exercise Group; Telehealth Exercise Group

SUMMARY:
Smoking can damage lung functions as a result of high carbon monoxide and low hemoglobin oxygen carrying capacity in the blood. Smoking between young people continues to increase, which can cause respiratory function problems and lung diseases at an early age. In the studies, it has been seen that smoking may reduce the oppression and exercise ability.

DETAILED DESCRIPTION:
Students who voluntarily accept participation in the study and sign the illuminated consent form, pulmonary status, gender, age, and body mass index to question data such as demographic data form, nicotine dependence levels Fagerstrom nicotine dependence scale, international physical activity scale (IPAQ), and Beck depression scale will be used. Then the respiratory function test will be evaluated with respiratory parameters and a 6-minute walking test. All evaluations made at the beginning of the study will be applied three times after the 8-week exercise program and the first month of control. First of all, the students will be grouped according to nicotine dependence levels, and exercise groups will be randomized according to each addiction level. Groups to be formed: Group 1: face-to-face exercise group; Group 2: online (telesağlık) exercise group; Group 3: control group.

ELIGIBILITY:
Inclusion Criteria:

* Signing the illuminated consent form,
* To be smoking at least 1 cigarette a day for the last 6 months,
* Not having orthopedic or neurological findings that can prevent the exercises included in the study,
* To have low-medium level physical activity level,
* Not to have any lower respiratory infection in the last 3 months.

Exclusion Criteria:

* To the exercise sessions to be held on time and not to arrive regularly

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (Short) | Evaluation should be carried out before the start of treatment and 8 weeks after treatment.
  It contains questions about the physical time spent in the last 7 days to learn about the physical activities of people in daily life. Metabolic equivalent (met) method was used to determine the level of physical activity. Standard Met values have been created for these activities. The daily and weekly physical activity level of the individual will be calculated by using the metal values determined for severe physical activity, moderate severe physical activity, walking and sitting.
Six-Minute Walk Test | Evaluation should be carried out before the start of treatment and 8 weeks after treatment.
  It is a widely used test for evaluating the functional capacity of individuals. Individuals shall be requested to walk at normal walking speeds in a flat corridor of thirty meters long, with the start and end points determined for six minutes, and the distance in which the cases walk for six minutes shall be recorded in meters.
Scoring the Fagerstrom Test for Nicotine Dependence (FTND) | Evaluation should be carried out before the start of treatment and 8 weeks after treatment.
  It is used to measure nicotine addiction. Points obtained from the scale, nicotine addiction level 0-2 Points: Very low level of nicotine addiction 3-4 points: low level of nicotine addiction, 5 points: moderate nicotine addiction, 6-7 points: high level of nicotine addiction, 8-10 points 8-10 points : It is classified as a very high level of nicotine addiction
Beck's Depression Inventory (BDI) | Evaluation should be carried out before the start of treatment and 8 weeks after treatment.
  It is a scale applied to determine whether the person shows signs of depression. The scale consists of 21 items, and eleven items are divided into cognitions, two substances, two substances, five substances, physical symptoms, and one substance for individual symptoms. Each question is given to 0, 1, 2, or 3, and the patients are asked to choose the most appropriate one of these questions. A score between 0-63 is obtained. 0-9 no/minimal depression, 10-18 mild depression, 19-29 moderate depression, and 30-63 severe depression.
Lung Function Test | Evaluation should be carried out before the start of treatment and 8 weeks after treatment.
  It allows the measurement of spirometry and pulmonary functions and the determination of abnormalities in the respiratory system. Spirometry shows the values obtained by exhalation and inhalation of air volumes during compulsory maneuvers. The main spirometry parameters are vital capacity (VC), challenging vital capacity (FVC), challenging expiratory volume in the first second (Fev1), and these parameters (Fev1/VC, Fev1/FVC).

CONTACTS AND LOCATIONS:
Locations (1):
- Kirklareli University, Kırklareli, Kayalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uysal MA, Kadakal F, Karsidag C, Bayram NG, Uysal O, Yilmaz V. Fagerstrom test for nicotine dependence: reliability in a Turkish sample and factor analysis. Tuberk Toraks. 2004;52(2):115-21. PMID 15241694
- [Result] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Result] Fagerstrom KO, Schneider NG. Measuring nicotine dependence: a review of the Fagerstrom Tolerance Questionnaire. J Behav Med. 1989 Apr;12(2):159-82. doi: 10.1007/BF00846549. PMID 2668531